CLINICAL TRIAL: NCT04578015
Title: A Randomized Controlled Trial of Treatment of Bacterial Vaginosis in Late Third Trimester to Prevent Maternal Peripartum Infection
Brief Title: A Randomized Controlled Trial of Treatment of Bacterial Vaginosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After screening many patients for BV, it was determined that the rate of BV is less in our population that the 30% rate mentioned in the literature. It was determined that completing the study will not be feasible due to cost and time constraints.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kartik K Venkatesh, MD, PhD Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020H0476
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Bacterial Vaginoses
Keywords: Bacterial Vaginoses; Cesarean delivery; Surgical site infection; Endometritis; Infection; Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial; Surgical Wound Infection; Endometritis; Infections; Vaginitis | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metronidazole 500 mg (Active Comparator): Participants in this arm will receive metronidazole 500 mg twice daily, orally for 7 days
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): Participants in this arm will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole — Participants in this arm will receive metronidazole 500 mg twice daily, orally for 7 days
  Arms: Metronidazole 500 mg
Drug: Placebo — Participants in this arm will receive placebo
  Arms: Placebo

SUMMARY:
This is a double-blinded, placebo controlled, multi-center randomized trial of 482 pregnant women who are diagnosed with Bacterial Vaginosis (BV) in the late 3rd trimester (>34 weeks). During routine clinic visit after 34 weeks, prospective patients will be counseled about the study. Patients who agree to be enrolled, will sign informed consent. Following enrollment, patients will be screened for BV. Those patients who are BV positive by clinical diagnosis, will be randomized to receive either metronidazole 500 mg BID orally for 7 days or identically appearing placebo.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 to ≤50 years with the ability to give informed consent.
* Patients expected to have a vaginal delivery with no obstetric contraindication for vaginal delivery at time of screening.
* Diagnosed with bacterial BV per Amsel criteria at time of screening in clinic.
* Gestational age ≥ 35 weeks

Exclusion Criteria:

* Plan for elective cesarean delivery
* Allergy or contraindications to metronidazole
* Receipt of metronidazole or clindamycin on admission for delivery for other indications.
* Hemodialysis
* Severe liver dysfunction
* Patient reports BV to nurse or clinician provider at current clinic visit or has been treated for BV within the past 3 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metronidazole 500 mg | Placebo
Started | 8 | 8
Completed | 0 | 0
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Population: Baseline analysis population data was not obtained as participants assigned to the treatment and placebo group did not complete the study, and this study was terminated due to lack of participant enrollment before data could be collected. No baseline data was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronidazole 500 mg | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Evaluating Composite of Chorioamnionitis, Postpartum Endometritis, SSI, Wound Infection, or Other Post-cesarean Infections (Occurring Within 6 Weeks After Delivery)
Time Frame: Through study completion, approximately 9.5 months
Population: Study outcomes were not collected as no participants completed either the intervention or control study group. Participation was terminated before completion of the study.
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Evaluating Incidence of Individual Infections.
Description: Chorioamnionitis, endometritis, wound infection (including necrotizing fascitis), other infections including abscess, septic thrombosis, pneumonia, pyelonephritis and breast infection.
Time Frame: At the time of admission for labor trough study completion, approximately 9.5 months
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Evaluating Incidence of Maternal Death
Time Frame: After delivery through study completion, approximately 9.5 months
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Evaluating Incidence of Puerperal Fever.
Description: Temperature > 100.4 F at least twice 30 minutes apart, or once with the use of antipyretic, or ≥101 F once.
Time Frame: Through study completion, approximately 9.5 months
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Evaluating Incidence of Use of Resources.
Description: Hospital stay, postpartum clinic or emergency room visit within 4 weeks of delivery, need for imaging or other invasive procedures, postpartum antibiotic use.
Time Frame: Through study completion, approximately 9.5 months
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Evaluating Incidence of Adverse Events
Description: Allergic reactions (anaphylaxis, angioedema, skin rashes including Stevens Johnson and Toxic Epidermal necrolysis), GI symptoms (nausea, vomiting, diarrhea, constipation, ileus, etc)
Time Frame: Through study completion, approximately 9.5 months
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Evaluating Incidence of Suspected Sepsis for Newborns
Time Frame: Within 7 days of delivery
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Evaluating Incidence of Confirmed Sepsis for Newborns
Time Frame: Within 7 days of delivery
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Evaluating Incidence of Newborn Intensive Care Unit (NICU) Admission and Duration
Time Frame: After delivery through study completion, approximately 9.5 months
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Evaluating Incidence of Neonatal Morbidities
Time Frame: After delivery through study completion, approximately 9.5 months
Population: as for outcome 1
Arm/Group | Metronidazole 500 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study termination
Description: No adverse events were observed prior to termination of the study.
Arm/Group | Metronidazole 500 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT04578015/Prot_SAP_000.pdf